CLINICAL TRIAL: NCT01465490
Title: Monitoring and Feedback in Substance Abuse Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Treatment Research Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: Public Health Management Corporation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA021154; 5R01DA021154-03 (NIH)
Record Dates: First submitted 2011-11-01; First posted 2011-11-04 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Substance Abuse
Keywords: Monitoring; Feedback; Substance Abuse Treatment
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monitoring and Feedback Intervention (Experimental)
  Interventions: Behavioral: Monitoring and Feedback Intervention
- Treatment as usual (No Intervention)

INTERVENTIONS:
Behavioral: Monitoring and Feedback Intervention — Clients participate in standard treatment and complete the MMI weekly with their counselors at the beginning of each individual counseling session. Counselors have been trained to administer the MMI and will have access to the data to use during sessions.
  Arms: Monitoring and Feedback Intervention

SUMMARY:
This is a three-staged study to develop and evaluate a monitoring instrument and associated intervention, as follows:

Stage 1 - Develop and determine the reliability, validity, and sensitivity to change of a brief Multidimensional Monitoring Instrument (MMI) for clients in outpatient substance abuse treatment (SAT).

Stage 2 - Develop a Monitoring and Feedback Intervention (MFI) that uses the MMI. As part of this process, create a manual, training materials, and competence and adherence measures, and conduct a feasibility study within an outpatient SAT unit to refine the intervention and associated materials and measures.

Stage 3 - Conduct a randomized clinical trial (RCT) to determine the preliminary efficacy of the MFI compared to treatment as usual (TAU) for clients in outpatient SAT. In this pilot study, it is hypothesized that the MFI will positively impact the treatment process, and short-term, during treatment, outcomes.

DETAILED DESCRIPTION:
In Stage 1, 20 substance abuse treatment (SAT) professionals, including clinicians, supervisors, and administrators, will participate in clinical focus groups. Clinical focus group members will review and discuss the MMI, its potential uses, and specific strategies around its implementation. Also in Stage 1, 240 clients will participate in a formal psychometric evaluation study of the Multidimensional Monitoring Instrument (MMI). These participants will complete a study intake meeting, which will include providing locator information (to facilitate scheduling research appointments), a baseline ASI6, and the MMI. After this intake, participants will complete 5 additional MMIs during a 4-week period. At the one and two-month follow-up research meetings, participants will complete the ASI6 and provide specimens for urine drug screens (UDSs). To ensure adequate resource management, participants who leave treatment at the program will not be continued in the study. Participants who are incarcerated during the study will not be contacted while in custody.

In Stage 2, the Monitoring and Feedback Intervention (MFI), the MFI Manual, and associated training materials will be completed with expert consultation. Also in Stage 2, 35 clients will participate in the MFI Feasibility Study. They will complete a baseline ASI6, as well as brief research assessments at 1-month post study intake and 2 months later (i.e., at the conclusion of their participation). Client participants will also provide specimens for UDSs. Clients will complete the MMI with their counselors on a regular basis, about weekly. Five randomly selected counselors will also participate in the Feasibility Study. They will meet with research staff for training and to periodically complete questionnaires/interviews. All individual counseling sessions will be recorded using a digital voice recorder.

During Stage 3, 112 clients will participate in a randomized clinical trial (RCT) of the intervention (MFI). These participants will complete a baseline ASI6, as well as brief research assessments at 1-month post study intake and 2 months later (i.e., at the conclusion of their participation). They will also provide samples for UDSs. Clients will be randomized so that one-half will receive treatment as usual (TAU; with the exception that counseling sessions will be digitally recorded), and one-half will receive MFI. Clients in the MFI group will participate in standard treatment and complete the MMI weekly with their counselors at the beginning of each individual counseling session. Also, a total of 8 counselors will be randomly selected to participate. They will be randomized so that 4 will provide TAU, and 4 will provide MFI. All counselors will meet with research staff for training and to periodically complete questionnaires/interviews. All individual counseling sessions will be recorded using a digital voice recorder.

ELIGIBILITY:
Inclusion Criteria:

* Client receiving intensive outpatient treatment at participating program
* Counselor employed by participating program

Exclusion Criteria:

* Client unable to speak English
* Client too cognitively impaired to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Treatment attendance | 3 months after consent
  Client participant's treatment attendance is obtained from treatment program clinical record.

SECONDARY OUTCOMES:
Urine screen results | 3 months after consent
  Client participant's urine screen results are obtained from treatment program clinical record.
Discharge status | 3 months after consent
  Client participant's discharge status is obtained from treatment program clinical record.
Discharge date | 3 months after consent
  Client participant's discharge date is obtained from treatment program clinical record.

CONTACTS AND LOCATIONS:
Overall Officials: John S Cacciola, Ph.D., Principal Investigator — Treatment Research Institute
Locations (4):
- United States (4):
  - Rehab After Work, Philadelphia, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Sobriety Through Outpatient, Philadelphia, Pennsylvania
  - Jefferson Intensive Outpatient, Philadelphia, Pennsylvania